CLINICAL TRIAL: NCT06092541
Title: Comparison of Efficacy Between Nitrous Oxide (n2o) Analgesia and Pericervical Analgesia in Outpatient Operative Hysteroscopy With Miniresector: a Randomized Clinical Pilot Study
Brief Title: Pericervical Analgesia Versus Analesia With Nitrous Oxide (N2O) in Outpatien Operative Hysteroscopy With Miniresector
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale degli Infermi di Biella (Other)
Responsible Party: Principal Investigator, Bianca Masturzo, Head of Obstetrics and Gynecology, Ospedale degli Infermi di Biella
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE 130/2023
Record Dates: First submitted 2023-10-04; First posted 2023-10-23 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Hysteroscopy
Keywords: hysteroscopy; pain control; pericervical anesthesia; nitrous oxide
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized clinical pilot study with masked third-party assessment. Patients will be assigned to the two groups (pericervical analgesia / nitrous oxide) through the sealed envelope method.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients, in the database, will be identified as group A and B; Once the study and the compilation of the database have been completed, this will be delivered to the results evaluation team which will therefore be blinded, not being able to recognize whether group A and B belong to control or intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: pericervical anesthesia (Experimental): Intervention group: pericervical anesthesia
  Interventions: Drug: Intervention Group: pericervical anesthesia
- Control group: nitrous oxide anesthesia (Active Comparator): Control group: nitrous oxide anesthesia
  Interventions: Other: Nitroux Oxide anesthesia

INTERVENTIONS:
Drug: Intervention Group: pericervical anesthesia — Patients assigned to the Intervention Group will receive Pericervical anesthesia before performing Hysteroscopy.
  Specifically, for the administration of pericervical analgesia, Mepivacaine/Lidocaine 1.5% 10/15 ml (max dose 7 mg/kg) will be used and pericervical infiltration will be performed at 0.5 cm depth at 3 and 9 hours.
  Other Names: Pericervical Anesthesia
  Arms: Intervention group: pericervical anesthesia
Other: Nitroux Oxide anesthesia — Patients assigned to the Control Group will receive Nitrous Oxide anesthesia before hysteroscopy
  Other Names: N2O2 Anesthesia
  Arms: Control group: nitrous oxide anesthesia

SUMMARY:
This research will have the aim of evaluating and comparing the effectiveness of two methods (analgesia with nitrous oxide and pericervical analgesia, excluding the use of paracervical block due to the increased risk of complications reported in the literature in the control of pain caused during Outpatient Operative Hysteroscopy maneuvers with Miniresector.

DETAILED DESCRIPTION:
Pain is the primary cause of hysteroscopy failure. It can be attributed to multiple causes, such as manipulation of the cervical canal , uterine distention due to the liquid distension media used during the procedure , operating procedures on the endometrium (as a possible cause of uterine contraction) , until the release of prostaglandins following manipulation of the cervix and uterine distension.

There are few studies in the literature that have compared the various methods of pain control during the hysteroscopic examination. Among these, Ahmad et al., for example, compared the use of the paracervical block and inhalation anesthesia during hysteroscopy: although both proved to be effective in controlling pain, the paracervical block was associated with a greater number of complications. More recently, Solano et al. they defined how the administration of nitrous oxide was equally effective (but with many more advantages) to the paracervical block with 1% lidocaine in controlling pain during hysteroscopy performed using the Bettocchi hysteroscope.

However, for the purposes of this research it is important to take two aspects into consideration:

* all the studies in the literature that compared the various pain control methods during hysteroscopy were conducted using the Bettocchi Hysteroscope and not the Miniresector;
* more in detail, there are no studies comparing the use of nitrous oxide and pericervical analgesia during outpatient operative hysteroscopy with miniresector.

Objective This clinical trial will have the aim of evaluating and comparing the effectiveness of two methods (analgesia with nitrous oxide and pericervical analgesia, excluding the use of paracervical block due to the increased risk of complications reported in the literature1) in the control of pain caused during Outpatient Operative Hysteroscopy maneuvers with Miniresector.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous or primiparous women (a previous Spontaneous Vaginal Birth -PS- or a previous Cesarean Section -TC- the latter comparable to nulliparous women as no previous cervical dilation -)
* age between 25 and 50 years

Exclusion Criteria:

* age < 25 or > 50 years
* multiparity
* positive history of previous operations on the cervical canal (e.g. conization)

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Rate of pain, measured through the Visual Analog Scale 1 (no pain) to 10 (worse pain) using Pericervical Analgesia versus Analgesia with Nitrous Oxide in outpatient hysteroscopic surgery with Miniresector | 6 months
  Change From Baseline in Pain Scores on the Visual Analog Scale -VAS- using Pericervical Analgesia versus Analgesia with Nitrous Oxide in outpatient hysteroscopic surgery with Miniresector

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Masturzo, MD PhD, Principal Investigator — Ospedale degli Infermi Biella
Locations (1):
- Ospedale degli Infermi, Biella, Italy

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, CSR
Time Frame: At the end of the study, for 6 months from the 1st may 2024 to 1st November 2024
Access Criteria: Participants centers

REFERENCES:
- [Background] Dealberti D, Riboni F, Prigione S, Pisani C, Rovetta E, Montella F, Garuti G. New mini-resectoscope: analysis of preliminary quality results in outpatient hysteroscopic polypectomy. Arch Gynecol Obstet. 2013 Aug;288(2):349-53. doi: 10.1007/s00404-013-2754-7. Epub 2013 Feb 16. PMID 23417150
- [Background] Ahmad G, Saluja S, O'Flynn H, Sorrentino A, Leach D, Watson A. Pain relief for outpatient hysteroscopy. Cochrane Database Syst Rev. 2017 Oct 5;(10)(10):CD007710. doi: 10.1002/14651858.CD007710.pub3. PMID 35611933
- [Background] Meyer L, Moore J, McMillan L. Outpatient Hysteroscopy in the Management of Abnormal Vaginal Bleeding. J Am Assoc Gynecol Laparosc. 1996 Aug;3(4, Supplement):S30-1. doi: 10.1016/s1074-3804(96)80239-8. PMID 9074183
- [Background] Zupi E, Luciano AA, Marconi D, Valli E, Patrizi G, Romanini C. The use of topical anesthesia in diagnostic hysteroscopy and endometrial biopsy. J Am Assoc Gynecol Laparosc. 1994 May;1(3):249-52. doi: 10.1016/s1074-3804(05)81018-7. PMID 9050495
- [Background] Solano Calvo JA, Del Valle Rubido C, Rodriguez-Miguel A, de Abajo FJ, Delgado Espeja JJ, Gonzalez Hinojosa J, Fernandez Munoz L, Zapico Goni A. Nitrous oxide versus lidocaine versus no analgesic for in-office hysteroscopy: a randomised clinical trial. BJOG. 2021 Jul;128(8):1364-1372. doi: 10.1111/1471-0528.16657. Epub 2021 Mar 9. PMID 33528862
- [Background] Del Valle Rubido C, Solano Calvo JA, Rodriguez Miguel A, Delgado Espeja JJ, Gonzalez Hinojosa J, Zapico Goni A. Inhalation analgesia with nitrous oxide versus other analgesic techniques in hysteroscopic polypectomy: a pilot study. J Minim Invasive Gynecol. 2015 May-Jun;22(4):595-600. doi: 10.1016/j.jmig.2015.01.005. Epub 2015 Jan 14. PMID 25596171
- [Background] De Silva PM, Carnegy A, Graham C, Smith PP, Clark TJ. Conscious sedation for office hysteroscopy: A systematic review and meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2021 Nov;266:89-98. doi: 10.1016/j.ejogrb.2021.09.001. Epub 2021 Sep 3. PMID 34600190
- [Background] Vitale SG, Alonso Pacheco L, Haimovich S, Riemma G, De Angelis MC, Carugno J, Lasmar RB, Di Spiezio Sardo A. Pain management for in-office hysteroscopy. A practical decalogue for the operator. J Gynecol Obstet Hum Reprod. 2021 Jan;50(1):101976. doi: 10.1016/j.jogoh.2020.101976. Epub 2020 Nov 6. PMID 33166706
- [Background] De Silva PM, Mahmud A, Smith PP, Clark TJ. Analgesia for Office Hysteroscopy: A Systematic Review and Meta-analysis. J Minim Invasive Gynecol. 2020 Jul-Aug;27(5):1034-1047. doi: 10.1016/j.jmig.2020.01.008. Epub 2020 Jan 23. PMID 31982584
- [Background] Schneider EN, Riley R, Espey E, Mishra SI, Singh RH. Nitrous oxide for pain management during in-office hysteroscopic sterilization: a randomized controlled trial. Contraception. 2017 Mar;95(3):239-244. doi: 10.1016/j.contraception.2016.09.006. Epub 2016 Sep 9. PMID 27621048
- [Background] Munro MG, Brooks PG. Use of local anesthesia for office diagnostic and operative hysteroscopy. J Minim Invasive Gynecol. 2010 Nov-Dec;17(6):709-18. doi: 10.1016/j.jmig.2010.07.009. PMID 20955982
- [Background] Keyhan S, Munro MG. Office diagnostic and operative hysteroscopy using local anesthesia only: an analysis of patient reported pain and other procedural outcomes. J Minim Invasive Gynecol. 2014 Sep-Oct;21(5):791-8. doi: 10.1016/j.jmig.2014.03.006. Epub 2014 Mar 25. PMID 24681061
- [Background] De Iaco P, Marabini A, Stefanetti M, Del Vecchio C, Bovicelli L. Acceptability and pain of outpatient hysteroscopy. J Am Assoc Gynecol Laparosc. 2000 Feb;7(1):71-5. doi: 10.1016/s1074-3804(00)80012-2. PMID 10648742
- [Background] The Use of Hysteroscopy for the Diagnosis and Treatment of Intrauterine Pathology: ACOG Committee Opinion, Number 800. Obstet Gynecol. 2020 Mar;135(3):e138-e148. doi: 10.1097/AOG.0000000000003712. PMID 32080054
- [Background] Ahlbom A. Modern Epidemiology, 4th edition. TL Lash, TJ VanderWeele, S Haneuse, KJ Rothman. Wolters Kluwer, 2021. Eur J Epidemiol. 2021 Aug;36(8):767-768. doi: 10.1007/s10654-021-00778-w. Epub 2021 Jul 3. No abstract available. PMID 34216355